CLINICAL TRIAL: NCT06364254
Title: The Effects of CBD on 2 Mile Run Time Trial Performance, GI Distress, and Anxiety in Moderately Active Females
Brief Title: Effects of CBD on 2 Mile Run Time Trial Performance
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Northern Colorado (Other)
Responsible Party: Principal Investigator, Laura Stewart, Professor, University of Northern Colorado
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 2311054791
Record Dates: First submitted 2024-03-08; First posted 2024-04-15 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Cannabidiol
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Cannabidiol capsules 2 hours prior to 2 mile run.
  Interventions: Dietary Supplement: Cannabidiol Capsules
- Placebo (Placebo Comparator): Placebo capsules 2 hours prior to 2 mile run.
  Interventions: Dietary Supplement: Cannabidiol Capsules

INTERVENTIONS:
Dietary Supplement: Cannabidiol Capsules — 300 mg of cannabidiol administered 2 hours before 2 mile run

SUMMARY:
Individuals who engage in endurance events tend to experience higher levels of stress within the body, mind, and gut, that often lead to impairment of performance. Based on previous studies, CBD has the potential relieve gut distress, and reduce pre-race anxiety thus resulting in an improvement in sport performance. Given the current research on the use of CBD in active individuals, the aim of this pilot study is to explore the effects of CBD compared to a placebo on anxiety, GI distress and a 2-mile running performance in a moderately active population identifying as female.

DETAILED DESCRIPTION:
This study will recruit moderately active, healthy individuals (N=30) who identify as female between the ages of 18-40 years who have some running experience and are running at least 2 miles, 2 times per week. This will be a cross over study, so each participant will be their own control, receiving either the placebo and CBD on two separate occasions. The females recruited will report to the Exercise Physiology lab in Gunter Hall on the University of Northern Colorado's campus for testing a total of two times.

The first visit will include initial paperwork such as the informed consent, physical activity readiness questionnaire (PARQ), Menstrual Cycle Questionnaire and a screening to determine current activity levels, uses CBD, THC and any other legal drugs/medications. This first interaction allows study staff to ensure that qualify to take part in the study.

After informed consent is obtained, the participant will be given either the placebo or CBD capsule with a controlled higher fat food (88 Acres protein bar) 2 hours before the testing protocol along. Once the CBD capsule or placebo is taken, participants will complete caffeine consumption, exercise and running questionnaires which will be administered on a tablet with study staff after 1.5 hours or waiting.

During the first visit, individuals will stay for a standardized period (2 hours) before doing a urine analysis to determine hydration status and taking v lactate, and heart rate variability. Current anxiety symptoms will also be evaluated

Once baseline measurements obtained, individuals will then be instructed to run 2 miles a treadmill as fast as possible. Lactate will be monitored three times during the test (.50 mile mark, halfway point (1 mile) and just before finishing the time trial run at the 1.98 mile mark). All participants will be taken through a 30-minute cool down period walking 2.5 mph on the treadmill while having lactate measured every 5, 10, 15, and 30 minutes post finishing. Finish time, GI distress questionnaire, and overall feelings will be recorded post finish of the 2 mile time trial.

Participants will be given a 25-30 day time between visits 1 and 2 to ensure exercise during the same menstrual cycle phase (hormone cycle) for those that are cycling. During the second and final visit, participants will undergo the same procedure, however, will be given the opposite oral administration from the first visit (either placebo or CBD).

ELIGIBILITY:
Inclusion Criteria:

* Running at least 2 miles 2 times per week.

Exclusion Criteria:

* Current diagnosis of a chronic disease or serious mental health disorder.
* Current or use of cannabis or cannabis products within the past 4 weeks
* Currently in perimenopause or menopause, transgender female not undergoing hormone treatment (estrogen)
* Having any underlying health concerns or have any current injuries that can be worsened with exercise

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals identifying as female.
Enrollment: 30 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Time Trial Times | 10-25 minutes
  Time to run 2 miles on an indoor treadmill
Difference in Anxiety Measured with the State Trait Anxiety Inventory | 5 minutes
  This questionnaire will be administered just before each run to assess the individual's current anxiety symptoms.The State-Trait Anxiety Inventory (STAI) consists of 20 items aimed at evaluating trait anxiety and 20 for state anxiety. All items are rated on a 4-point scale (e.g., from "Not at all" to "Very much so"). Higher scores suggest elevated anxiety.
Difference in Blood Lactate Concentrations | 45 minutes
  Blood lactate will be measured just before the time trial, 3 minutes after the start of the run, after 1 mile and 1.98 miles of running and after 5, 10, 15, and 30 minutes of walking recovery. Higher lactate concentrations are associated with more effort during exercise and a slower recovery from exercise.
Difference in Gastrointestinal Distress | 5 minutes
  This questionnaire consists of 12 questions related to distress symptoms. Responses are absent, mild, moderate, severe. The higher the score, the more GI distress is present. This assessment will be completed after the 2 mile run.
Different in Heart Rate Variability | 5 minutes
  The root mean square successive difference method will be used with the 10 second electrocardiogram reading. Higher heart rate variability is associated with better health.

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Northern Colorado, Greeley, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided